CLINICAL TRIAL: NCT03850964
Title: A Phase II/III Randomized, Placebo Controlled, Double Blind Study to Evaluate the Effects of up to 24 Weeks of Low Dose Pazopanib on Hereditary Hemorrhagic Telangiectasia Related Epistaxis and Anemia
Brief Title: Effects of Pazopanib on Hereditary Hemorrhagic Telangiectasia Related Epistaxis and Anemia (Paz)
Acronym: Paz
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cure HHT (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HT2; CDMRP-PR203473 (Other Grant/Funding Number: US Department of Defense USAMRAA); 1R01FD006840-01A1 (FDA)
Record Dates: First submitted 2019-02-12; First posted 2019-02-22 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2024-11

CONDITIONS: Hereditary Hemorrhagic Telangiectasia; Epistaxis; Anemia; Nosebleed; HHT
Keywords: Osler-Weber-Rendu; Hereditary Hemorrhagic Telangiectasia; Patient Reported Outcome; HHT; Anemia; Nosebleed; Epistaxis
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Epistaxis; Anemia | interventions — pazopanib; Cellulose

STUDY DESIGN:
Intervention Model Description: After at least a 6-week baseline period, participants will be assigned low dose pazopanib (150 mg) or placebo.
  At the termination of the 24-week Efficacy study participants will be provided the option to advance into an open label extension program including 24 weeks of treatment, followed by a 12-week non-drug follow up period. The extension would be on active drug, but otherwise blinded to the dose provided in the primary trial.
  This decision to continue into the extension will be based on a physician-participant discussion of any efficacy and safety concerns at week 24. A decision would be reached whether to proceed into the extension study and whether to consider a dose modification. A top dose of 150 mg will be maintained.
  After the extension, a 12 week follow-up time period will continue assessments to define maintenance of effect, and/ or relapse.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Project Manager in operation will also be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Part B (Severe Anemia) Pazopanib - 150 mg (Active Comparator): 150 mg pazopanib oral capsules (six 25 mg placebo capsules daily).
  Interventions: Drug: Pazopanib
- Part B (Severe Anemia) Placebo (Placebo Comparator): Placebo oral capsules (six 25 mg placebo capsules daily).
  Interventions: Drug: Placebo oral capsule
- Part B (Severe Epistaxis) Pazopanib - 150 mg (Active Comparator): Pazopanib 150 mg oral daily dosing (six 25 mg Pazopanib capsules).
  Interventions: Drug: Pazopanib
- Part B (Severe Epistaxis) Placebo (Placebo Comparator): Placebo oral capsules (six 25 mg placebo capsules daily).
  Interventions: Drug: Placebo oral capsule
- Part C Pazopanib - 150 mg (Experimental): Pazopanib 150 mg oral daily dosing (six 25 mg Pazopanib capsules).
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib — gel capsule, with 25mg-similar fills
  Other Names: Votrient
  Arms: Part B (Severe Anemia) Pazopanib - 150 mg; Part B (Severe Epistaxis) Pazopanib - 150 mg; Part C Pazopanib - 150 mg
Drug: Placebo oral capsule — identical gel capsule without active pharmaceutical ingredient
  Other Names: cellulose capsule
  Arms: Part B (Severe Anemia) Placebo; Part B (Severe Epistaxis) Placebo

SUMMARY:
During the Efficacy Study (Part B), the investigators will study whether Pazopanib, taken daily for 24 weeks, will reduce the severity of nose bleeds in patients with hereditary hemorrhagic telangiectasia (HHT). Patients will either be provided active drug or a placebo [sugar - inactive pill], and be tested for nose bleed severity throughout the trial, including particularly nose bleed duration. Investigators will also test for blood loss, as well as for safety. This study is funded by the US Department of Defense USAMRAA and FDA/OOPD.

DETAILED DESCRIPTION:
Now that a single dose pharmacokinetics (PK) study (Part A) has been completed to properly establish similar exposure with the prior pilot 50mg tablet, a double blind, placebo controlled study will follow (Part B), which proposes to define primarily the value of low dose (150 mg) Pazopanib on nose bleed duration, in the context of assessing perceived nose bleed severity.

After a patient completes Part B of the study, the patient will be invited to take part in an Extension Study (Part C) in which the patient will be provided with active drug equal to the dose they were assigned in Part B. All patients in Part C will receive active drug for 24 weeks. Part C will further assess the effects of Pazopanib on the severity of nose bleeds in patients with HHT and also support safety and efficacy elements.

After the patient completes their treatment period (either Part B or Parts B and C), a 12 week follow-up period will follow to support safety and efficacy elements. Secondary endpoints will be assessed, including ongoing blood loss, use of iron and blood products, quality of life, and drug safety.

ELIGIBILITY:
Part B

Inclusion Criteria (all of the following are necessary):

* A definite or probable diagnosis of hereditary hemorrhagic telangiectasia (HHT):

  1. Definite clinical HHT defined as having at least 3 of the following criteria:

     * Spontaneous and recurrent epistaxis.
     * Multiple telangiectasias at characteristic sites: lips, oral cavity, fingers, nose.
     * Visceral lesions: GI telangiectasia, pulmonary, hepatic, cerebral or spinal AVMs.
     * A first degree relative with HHT according to these criteria.
  2. OR a definite diagnosis of HHT based on a pathogenic genetic mutation for HHT.
  3. OR probable HHT based on having 2 of the above criteria with high clinical suspicion of HHT.
* Stable IV iron use and/or blood transfusions stable for 12 weeks prior to test product initiation.
* Must agree not to undergo cautery of nasal telangiectasias or to start new therapies for HHT while on study.
* Women of childbearing potential must agree to abstinence or to use an acceptable double method contraception until 4 weeks after drug termination. Pregnancy testing will be done throughout the trial.
* Men are mandated to use condoms.
* Capable of giving signed informed consent.
* Able and willing to return for outpatient visits at the protocol specified intervals.
* Able and willing to complete blood pressure monitoring at home.
* Able and willing to complete daily patient reported outcome measurements at home.
* Must meet all of the inclusion criteria for either:

Severe Anemia Cohort:

i. Anemia mainly due to HHT (in the judgment of the PI) with average Hgb <10 g/dL regardless of gender (average of at least three measures during screening and run in).

ii. Epistaxis averaging at least 5 min/week over the six-week baseline and is generally stable in the clinical judgement of the investigator.

Severe Epistaxis Cohort:

i. Anemia mainly due to HHT (in the judgment of the PI) with Hgb <12 g/dL in women or <13 g/dL in men (average of at least three measures during screening and run in).

ii. Epistaxis averaging at least 20 min/week over the six-week baseline and is generally stable in the clinical judgement of the investigator.

Part B

Exclusion Criteria:

* Participant has known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to pazopanib that in the opinion of the investigator contradicts their participation.
* Currently has incompletely treated cerebral arterio-venous malformations (AVMs) or cerebral arteriovenous fistulas (AVFs) that are symptomatic or have high-risk features detected on either MRI/MRA or digital subtraction angiography. High-risk features include: microhemorrhage seen on MRI; feeding artery aneurysm, nidus aneurysm or venous outflow stenosis seen on MRA, CTA, or catheter angiography. Non-shunting vascular brain lesions such as capillary vascular malformations, telangiectasias, and cavernous malformations are not an exclusion criterion. (Note: MRI scan does not need to be repeated at screening if AVMs and AVFs were absent on a scan at age ≥18 years).
* Currently has perfused pulmonary AVMs with feeding artery diameter ≥ 3mm.
* Known significant bleeding sources other than nasal or gastrointestinal.
* Systemic use of a potent VEGF inhibitor (e.g., direct inhibitors of VEGF-receptor signaling such as sunitinib) in the 4 weeks prior to enrollment. Systemic use of bevacizumab in the 6 weeks prior to enrollment due to its longer half-life.
* Active and recent onset of clinically significant diarrhea.
* Current or recent (in the last 5 years) malignancies (except non-melanoma skin cancers)
* Participant has had major surgery (e.g. surgical ligation of an AVM) or trauma within 28 days or had minor surgical procedures (e.g. central venous access line removal) within 7 days prior to dosing, the latter representing a recent wound, fracture or ulcer
* Participant has a planned surgery during periods of active treatment and 6 weeks of follow up; case by case evaluation if PI desires inclusion with medical monitor agreement.
* Participant has clinically significant gastrointestinal abnormalities (other than hereditary hemorrhagic telangiectasia related vascular lesions).
* Participant during the 6 months prior to first dose of study drug has a history of cerebrovascular accident (including transient ischemic attacks), pulmonary embolism, untreated deep vein thrombosis (DVT), myocardial infarction, or any other thrombotic event.
* Presence of intrinsic heart disease as evidenced by any of the following: Echo derived left ventricular ejection fraction < 45%; Unstable obstructive CAD; history of MI, CABG, or PCI in the last 6 months; Infiltrative and/or restrictive cardiomyopathies; Significant pericardial disease; or clinical heart failure with more than moderate mitral valve or aortic valve disease. In the absence of clinical heart failure, EKG abnormalities, or known cardiac functional disease (e.g., MI or cardiomyopathy), a previous echo during adulthood is adequate. If there is history for coronary disease or cardiomyopathy, an echo in the past 5 years will be adequate for screening. If the patient has current clinical heart failure, a recent cardiac event in last 5 yrs, or a cardiac event since the most recent echo, an echo in the past 6 months will be necessary for screening. Clinical heart failure due to liver AVM or anemia, and not associated with the above findings (with an EF >=45%) will be eligible for enrollment.
* Unable or unwilling to discontinue use of prohibited medications list in Section 6.5.2 for at least 14 days or 5 half-lives of a drug (whichever is longer) prior to the randomization and for the duration of the study.
* The participant has participated in a clinical trial and has received an investigational product within the following time period prior to the start of randomization: 4 weeks, 4 half-lives or the duration of the biological effect of the investigational product (whichever is longer).
* QT corrected interval >450 msec for men or >460 msec for women, based on averaged QT corrected interval values of triplicate ECGs obtained over a brief recording period.

  * History of familial prolonged QT.
  * Any concomitant medication which is known to prolong QT.
* Average baseline hemoglobin <6 g/dL.
* Platelets < 75x10^9 /L.
* International normalized ratio (INR) > 1.5x ULN or activated partial thromboplastin time (aPTT) > 1.5x ULN (unless due to known concurrent medications, e.g. warfarin).
* Alanine Transaminase (ALT) >2 x upper limit of normal.
* Bilirubin >1.5x upper limit of normal (isolated bilirubin >1.5x upper limit of normal is acceptable if bilirubin is fractionated and direct bilirubin < 35%).
* Participant has poorly controlled hypertension [defined as systolic blood pressure (SBP) ≥ 140 mmHg or diastolic blood pressure (DBP) ≥ 90 mmHg]. If BP is poorly controlled at screen visit, initiation or adjustment of antihypertensive medication(s) is permitted during the run-in period prior to randomization. Prior to randomization, blood pressure must be assessed three times and the mean SBP/DBP must be < 140/90 mmHg in order for a patient to be randomized.
* Substantive renal disease (eGFR <30 mL/min/1.73m2calculated using the Cockcroft-Gault formula)
* Echo derived left ventricular ejection fraction < 45%.
* Thyroid stimulating hormone (TSH) > 1.5 x upper limit of normal.
* Urine protein to creatinine ratio > 0.4.
* Neutrophil count <1000 /mm^3.

Part C Eligibility

All patients who completed Part B will be eligible for Part C unless significant safety concerns have been raised.

Participants must be able and willing to sign the Extension ICF.

Neither the Study Doctor or the participant will be informed of which drug (active or placebo) received during Part B.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in epistaxis duration in minutes | Average duration in weeks 19-24 (last 6 weeks of blinded phase) versus baseline.
  >=50% decrease in the duration of epistaxis in the 150 mg pazopanib arm versus the placebo arm (moderate and severe cohorts combined)
Hemoglobin Response rate increase in hemoglobin | Average duration in weeks 19-24 (last 6 weeks of blinded phase) versus baseline.
  Increase in hemoglobin by ≥ 2 g/dl in the 150 mg pazopanib arm versus the placebo arm (moderate and severe cohorts combined)

SECONDARY OUTCOMES:
Achievement of meaningful improvement in epistaxis for HHT patients | Baseline [screening, run-in and 0 time points] and week 24.
  Compare patients reported being bothered by epistaxis at baseline and report not bothered at week 24
Percent change in blood transfusion rate in the Severe Cohort | Baseline, and weeks 13-24
  Reduction in RBC transfusion rate by at least one unit
Assess the safety of up to 24 and 48 weeks of treatment of pazopanib | 1st dose of intervention until Weeks 24 and 48
  * AEs; absolute values and changes over time of hematology, clinical chemistry, urinalysis, blood pressure, and heart rate.
  * Physical exam, leg and abdominal evaluations, and CNS symptoms.
  * ECG parameters (PR, QRS, QT, QTc intervals) in addition to cardiac echocardiogram to evaluate LV function from pre-dose values in at-risk patients (baseline EF <50)
Assess pharmacokinetics and pharmacodynamics (PK/PD) of treatment | Weeks 12, 24, 36 and 48
  * Cτ, data permitting
  * Graphical exploration of PK/PD relationships between pazopanib and selected PD endpoints
Establish comparability of endpoint outcomes for each hemoglobin stratification | Baseline, Weeks 19-24, Week 48
  Trends for primary endpoint in severe (hemoglobin (<9.5 g/dl) and moderate (9.5-10.9 g/dl) groups.

OTHER OUTCOMES:
Assess effects of up to 24 weeks of pazopanib treatment on epistaxis duration | Baseline and weeks 19-24 of study.
  Decrease in Epistaxis duration by ≥50% averaged over weeks 19-24 versus baseline
Assess the effects of up to 24 weeks of pazopanib treatment on hemoglobin levels | Baseline and weeks 19-24 of study
  Increase in hemoglobin over the 24 weeks by 2g/dL of greater average over weeks 19-24 versus baseline (overall and stratified by hemoglobin)
Assess the effects of up to 24 weeks of pazopanib treatment on frequency of nose bleeds and speed of flow | Baseline and weeks 19-24 of study
  Establish percentage decrease in frequency of nose bleeds and speed of flow category improvement averaged over weeks 19-24 versus baseline
Change with pazopanib treatment for epistaxis frequency and speed of flow, and fatigue | Baseline, 12, 24, and 48 weeks
  Meaningful change quantities will be determined using domain-specific, patient-reported anchors focusing on importance and severity of change. Focus will be on change from baseline to 12, 24, and 48 weeks
Assess effects of up to 24 weeks of pazopanib treatment on epistaxis symptom elements | Baseline, 3-week dosing intervals over study
  Change in epistaxis: frequency, speed of flow, and epistaxis duration
Assess effect of up to 24 and 48 weeks of pazopanib treatment on level of epistaxis severity | Epistaxis severity - average of last 6 weeks of study compared to baseline 6 weeks; Change in ESS at 12, 24 and 48 weeks (versus baseline)
  * Change in level of epistaxis severity by at least one unit
  * Change in ESS by time
Change or reduction in iron supplementation for up to 48 weeks of treatment | Baseline, Week 19-24, Weeks 43-48
  IV and oral iron use (together and separately)
Effects of up to 48 weeks of pazopanib treatment on serum ferritin for all patients | Weeks 0, 12, 24, 36, and 48
  Serum ferritin levels
Effects of up to 48 weeks of pazopanib treatment on quality of life | Part B: Baseline, every 6 weeks; Part C: Baseline, every 12 weeks
  Changes in social and physical activity PROMIS self-reported questionnaire
Perceived benefits of up to 48 weeks of pazopanib treatment for reducing symptoms, specifically satisfaction | Week 24, 48 or early study termination visit
  Response to an exit interview at the last visit
Effects of up to 48 weeks of pazopanib treatment on cardiac function | Baseline, weeks 24 and 48
  * BNP protein levels in all patients
  * Echo, 6 min walk, and diuretic usage record in patients with clinical heart failure due to liver AVM
Examine the drug mechanism of pazopanib treatment | Baseline, Weeks 24 and 48
  Measure VEGFR2 serum values
Examine the role of genotype on response to pazopanib treatment | Weeks 24 and 48
  Epistaxis and hemoglobin outcomes stratified by genotype (Alk1, Endoglin, SMAD)

CONTACTS AND LOCATIONS:
Overall Officials: James Gossage, MD, Principal Investigator — Augusta University
Locations (11):
- United States (11):
  - University of California - Los Angeles, Los Angeles, California
  - University of Colorado, Denver, Colorado
  - Augusta University, Augusta, Georgia
  - John Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - University of North Carolina, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Texas - Southwestern, Dallas, Texas
  - University of Utah Medical Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
Over the first 18 months post study, the participating sites and PI's will produce primary and adjunct reports. After this period, study data will be posted on an available internet site for others to interrogate

REFERENCES:
- [Background] Faughnan ME, Gossage JR, Chakinala MM, Oh SP, Kasthuri R, Hughes CCW, McWilliams JP, Parambil JG, Vozoris N, Donaldson J, Paul G, Berry P, Sprecher DL. Pazopanib may reduce bleeding in hereditary hemorrhagic telangiectasia. Angiogenesis. 2019 Feb;22(1):145-155. doi: 10.1007/s10456-018-9646-1. Epub 2018 Sep 6. PMID 30191360
- [Background] Clark M, Berry P, Martin S, Harris N, Sprecher D, Olitsky S, Hoag JB. Nosebleeds in hereditary hemorrhagic telangiectasia: Development of a patient-completed daily eDiary. Laryngoscope Investig Otolaryngol. 2018 Nov 14;3(6):439-445. doi: 10.1002/lio2.211. eCollection 2018 Dec. PMID 30599027
- [Background] Parambil JG, Gossage JR, McCrae KR, Woodard TD, Menon KVN, Timmerman KL, Pederson DP, Sprecher DL, Al-Samkari H. Pazopanib for severe bleeding and transfusion-dependent anemia in hereditary hemorrhagic telangiectasia. Angiogenesis. 2022 Feb;25(1):87-97. doi: 10.1007/s10456-021-09807-4. Epub 2021 Jul 22. PMID 34292451